CLINICAL TRIAL: NCT04917692
Title: Empagliflozin in Adolescent Diabetes
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Not funded
Sponsor: Ohio State University (Other)
Collaborators: Diacomp (Unknown)
Responsible Party: Principal Investigator, Robert Hoffman, Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Empad
Record Dates: First submitted 2021-05-14; First posted 2021-06-08 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: type1diabetes
Keywords: type 1 diabetes; adolescents; cardiovascular risk; inflammation; complement; endothelial function; empagliflozin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Inflammation | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Single arm, open label intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- empagliflozin (Experimental): empagliflozin 2.5 mg daily
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — 2.5 mg daily
  Other Names: Jardiance

SUMMARY:
Empagliflozin, an inhibitor of the sodium glucose co-transporter 2 (SGLT2), reduces post-prandial glucose levels in adults with both type 2 and type 1 diabetes and importantly reduces both cardiovascular and renal complications in type 2 diabetes. In adults with type 1 diabetes empagliflozin improves endothelial function and vascular stiffness when used in conjunction with insulin. There is clear evidence that complications in type 1 diabetes have their origins during adolescents thus to reduce diabetic complications with adjunctive therapy, this age group must be studied. These studies will need to focus on the effects of these adjunctive agents on functional biomarkers for development of complications. This study is designed to develop pilot and feasibility data for a large scale trial of low dose empagliflozin, 2.5 mg daily, on biomarkers for the development of cardiovascular and renal complications in adolescents between 12 and 18 years of age. The investigators will specifically study the effects of 8 weeks of empagliflozin on:

1. Pre-and post-prandial inflammatory markers using high carbohydrate and high fat meals. Inflammatory markers to be measured include interleukin-6 (IL-6), tissue necrosing factor α (TNF-α), complement component C3 concentrations and skin advanced glycosylation endproducts (AGE).
2. Pre-and post-prandial vascular function including forearm vascular resistance, endothelial function and pulse wave velocity.
3. Microalbuminuria and pre- and post-prandial glomerular hyperfiltration, tubular injury and renal inflammation.

The investigators will, also, measure more traditional risk markers including blood pressure, hemoglobin A1c, and lipids. Eligible participants will have had diabetes for at least 1 year and not have other chronic medical illnesses or diabetes complications. Because of the risk of diabetic ketoacidosis (DKA) subjects must have a hemoglobin A1c level less than 9% and have no history of recurrent DKA or known insulin omission. This will be the first pilot study designed to explore primary endpoints regarding cardiovascular and renal disease rather than glucose control with empagliflozin therapy in adolescents with type 1 diabetes.

DETAILED DESCRIPTION:
This is an 8 week single arm trial on the effects of empagliflozin 2.5 mg in adolescents with type 1 diabetes for at least 1 year. Subjects will be studied in the Clinical Research Center of the Wexner Medical Center at the Ohio State University 3 times. Visit 0 will be the initial study visit and will involve obtaining informed consent and assent, taking a medical history and performing a physical examination. Over the next 2 weeks the subjects will be contacted by the investigators to adjust insulin doses.

Visit 1 will be the baseline visit. It will occur at 8AM after an overnight fast. Blood samples will be collected to measure inflammatory markers will be collected and vascular function will be tested. Subjects will then be given premeal insulin and a breakfast. Following this, additional blood samples and vascular function measurements will be taken at 30, 60, 90, and 120 minutes.

After completion of the tests home insulin doses will be reduced and the subjects will be given empagliflozin 2.5 mg daily to take at home for the next 8 weeks. They will be instructed regarding potential side effects including diabetic ketoacidosis and genital infections.

Subjects will be contacted regularly by the investigators during these 8 weeks to review home glucose monitoring and potential side effects. After completion of the 8 weeks Visit 2 will occur which will be identical Visit 1.

ELIGIBILITY:
Inclusion Criteria:

* Age: 12-18 years
* Clinical diagnosis of type 1 diabetes
* Duration of diabetes > 1 r
* Multiple daily injections or continuous subcutaneous insulin infusion.
* Home glucose testing 4 times per day or continuous glucose monitor.
* Hemoglobin A1c levels will be ≤ 10.5%
* History of adherence to insulin administration, carbohydrate counting.

Exclusion Criteria:

* Duration of type 1 diabetes for less than 1 year
* Medical conditions other than type 1 diabetes or treated hypothyroidism
* Medications other than insulin, levothyroxine or oral contraceptives for birth control
* Antihypertensive medications, lipid lowering medications, or anti-hyperglycemic agents other than insulin.
* Acute viral and bacterial illnesses are not exclusionary, but we will take a health history at baseline and at the time of any study visit and if a recent illness has occurred we will delay testing until the individual is symptom free for 1 week and off and treatment for the illness.
* Hospital admission for diabetic ketoacidosis in the last year

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Interleukin 6 | 8 weeks
  IL6 levels will be measured before and after high carbohydrate meal at the beginning and end of the 8 weeks
Glomerular filtration rate | 8 weeks
  Cystatin C levels will be used to calculate GFR before and after high carbohydrate meal at the beginning and end of the 8 weeks
Endothelial function | 8 weeks
  Percentage change in forearm vascular resistance following 5 min of arterial occlusion.
Number of episodes of diabetic ketoacidosis per patient | 8 weeks
  Frequency of diabetic ketoacidosis will be assessed through the 8 weeks

SECONDARY OUTCOMES:
Complement | 8 weeks
  Complement component C3 and C4 levels will be measured before and after high carbohydrate meal at the beginning and end of the 8 weeks
Lipids | 8 weeks
  Lipid levels will be measured before and after high carbohydrate meal at the beginning and end of the 8 weeks
Pulse wave velocity | 8 weeks
  Pulse wave velocity will be measured before and after high carbohydrate meal at the beginning and end of the 8 weeks
Number of episodes of hypoglycemia per patient | 8 weeks
  Frequency of hypoglycemia will be assessed over 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No